CLINICAL TRIAL: NCT06321614
Title: Self-supervised Learning for Classifying Bowel Obstruction on Upright Abdominal Radiography
Brief Title: Deep Learning in Classifying Bowel Obstruction Radiographs
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022098
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Digestive System Disease; Polyp of Colon; Bowel Disease
Keywords: Deep learning; Artificial intelligence; Machine learning
MeSH Terms: conditions — Digestive System Diseases; Colonic Polyps; Intestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with normal abdominal radiographs: patients with normal abdominal radiographs, which were confirmed by extra imaging examinations and clinical data. The imaging examinations comprised CT, magnetic resonance imaging (MRI) and colonoscopy in the subsequent 72 hours, while clinical data included recent hospital admission information and surgical operation notes.
- patients with small bowel obstruction radiographs: patients with small bowel obstruction radiographs, which were confirmed by extra imaging examinations and clinical data. The imaging examinations comprised CT, magnetic resonance imaging (MRI) and colonoscopy in the subsequent 72 hours, while clinical data included recent hospital admission information and surgical operation notes. In terms of location, small-bowel obstruction (SBO) involves the duodenum, jejunum, and ileum
- patients with large bowel obstruction radiographs: patients with large bowel obstruction radiographs, which were confirmed by extra imaging examinations and clinical data. The imaging examinations comprised CT, magnetic resonance imaging (MRI) and colonoscopy in the subsequent 72 hours, while clinical data included recent hospital admission information and surgical operation notes. In terms of location, large-bowel obstruction (SBO), involves the cecum, colon, and rectum.

SUMMARY:
Background: Accurate labeling of obstruction site on upright abdominal radiograph is a challenging task. The lack of ground truth leads to poor performance on supervised learning models. To address this issue, self-supervised learning (SSL) is proposed to classify normal, small bowel obstruction (SBO), and large bowel obstruction (LBO) radiographs using a few confirmed samples.

Methods: A few number of confirmed and a large number of unlabeled radiographs were categorized based on the ground truth. The SSL model was firstly trained on the unlabeled radiographs, and then fine-tuned on the confirmed radiographs. ResNet50 and VGG16 were used for the embedded base encoders, whose weights and parameters were adjusted during training process. Furthermore, it was tested on an independent dataset, compared with supervised learning models and human interpreters. Finally, the t-SNE and Grad-CAM were used to visualize the model's interpretation.

ELIGIBILITY:
Inclusion Criteria:

1. The hospital imaging system looked for plain abdominal standing films diagnosed as intestinal obstruction or normal between 2022 and 2024
2. Aged 18 to 80 years
3. The main complaint was gastrointestinal symptoms

Exclusion Criteria:

1. Image interference, fuzzy performance, difficult to distinguish
2. Non-gastrointestinal symptoms were the main complaint
3. Supine, prone, or lateral decubitus radiography
4. Paralytic obstruction, closed loop obstruction, et al

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants received upright abdominal radiographs were included in this study. They can be divided with participants with normal abdominal radiographs, participants with small bowel obstruction, and participants with large bowel obstruction. The study strictly follow the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and classification performance | 1 week
  Accuracy, Recall, Precision, F1-score and confusion matrix

SECONDARY OUTCOMES:
Visualized interpretation of the self-supervised model | 1 week
  Grad-CAM and t-SNE to visualize the interpretation of the SSL model

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, MD, Study Director — The First Affiliated Hospital of Soochow University
Locations (1):
- TheFirst Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Markogiannakis H, Messaris E, Dardamanis D, Pararas N, Tzertzemelis D, Giannopoulos P, Larentzakis A, Lagoudianakis E, Manouras A, Bramis I. Acute mechanical bowel obstruction: clinical presentation, etiology, management and outcome. World J Gastroenterol. 2007 Jan 21;13(3):432-7. doi: 10.3748/wjg.v13.i3.432. PMID 17230614
- [Result] Cheng PM, Tran KN, Whang G, Tejura TK. Refining Convolutional Neural Network Detection of Small-Bowel Obstruction in Conventional Radiography. AJR Am J Roentgenol. 2019 Feb;212(2):342-350. doi: 10.2214/AJR.18.20362. Epub 2018 Nov 26. PMID 30476452
- [Result] Kim DH, Wit H, Thurston M, Long M, Maskell GF, Strugnell MJ, Shetty D, Smith IM, Hollings NP. An artificial intelligence deep learning model for identification of small bowel obstruction on plain abdominal radiographs. Br J Radiol. 2021 Jun 1;94(1122):20201407. doi: 10.1259/bjr.20201407. Epub 2021 Apr 27. PMID 33904763
- [Result] Frager D. Intestinal obstruction role of CT. Gastroenterol Clin North Am. 2002 Sep;31(3):777-99. doi: 10.1016/s0889-8553(02)00026-2. PMID 12481731
- [Result] Cappell MS, Batke M. Mechanical obstruction of the small bowel and colon. Med Clin North Am. 2008 May;92(3):575-97, viii. doi: 10.1016/j.mcna.2008.01.003. PMID 18387377
- [Result] ten Broek RP, Strik C, Issa Y, Bleichrodt RP, van Goor H. Adhesiolysis-related morbidity in abdominal surgery. Ann Surg. 2013 Jul;258(1):98-106. doi: 10.1097/SLA.0b013e31826f4969. PMID 23013804
- [Result] Vanderbecq Q, Ardon R, De Reviers A, Ruppli C, Dallongeville A, Boulay-Coletta I, D'Assignies G, Zins M. Adhesion-related small bowel obstruction: deep learning for automatic transition-zone detection by CT. Insights Imaging. 2022 Jan 24;13(1):13. doi: 10.1186/s13244-021-01150-y. PMID 35072813
- [Result] Chen Y, Mancini M, Zhu X, Akata Z. Semi-Supervised and Unsupervised Deep Visual Learning: A Survey. IEEE Trans Pattern Anal Mach Intell. 2024 Mar;46(3):1327-1347. doi: 10.1109/TPAMI.2022.3201576. Epub 2024 Feb 6. PMID 36006881
- [Result] Li G, Togo R, Ogawa T, Haseyama M. Self-supervised learning for gastritis detection with gastric X-ray images. Int J Comput Assist Radiol Surg. 2023 Oct;18(10):1841-1848. doi: 10.1007/s11548-023-02891-5. Epub 2023 Apr 11. PMID 37040011